CLINICAL TRIAL: NCT07396857
Title: The Role of Endothelial-Derived Hyperpolarization Factors on 24-hr Blood Pressure Regulation Following a Bout of Prolonged Sitting
Brief Title: The Role of EDHFs on Blood Pressure Following a Bout of Prolonged Sitting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Principal Investigator, Myles William O'Brien, Assistant Professor, Université de Sherbrooke
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2025-7915
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Cardiovascular
Keywords: Arterial function; Sedentary time; Sex differences; Vasoactive substances
MeSH Terms: conditions — Sedentary Behavior | interventions — Fluconazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Males (Experimental)
  Interventions: Drug: Placebo; Drug: Fluconazole 150 mg
- Females (Experimental)
  Interventions: Drug: Placebo; Drug: Fluconazole 150 mg

INTERVENTIONS:
Drug: Placebo — Participants will take a placebo sugar pill before and after a bout of prolonged sitting as a control session.
Drug: Fluconazole 150 mg — Participants will take 150mg of fluconazole, an EDHF inhibitor before and after a bout of prolonged sitting.

SUMMARY:
Canadians spend most of their day in sedentary postures (i.e., sitting, lying, reclining). While the beneficial impacts of physical activity on the heart are well-established, less is known about the consequences during time spent in sedentary postures. Currently, we know that spending time in a bout of uninterrupted sitting disrupts blood pressure regulation. However, it is unknown if there are any 'carry over' effects following uninterrupted sitting bouts (i.e., over the next 24-hours). The release of chemicals from arteries controls how stiff or relaxed they are and is important for controlling blood pressure. This is especially true for arteries directly impacted by sitting (e.g., the popliteal artery behind the knee) and that send blood to the brain (e.g., the carotid artery). We have also established that endothelial-derived hyperpolarizing factors (EDHF, chemicals that relax the artery) are important for the relaxation of the artery the popliteal artery. However, we do not know if the effects of EDHFs on this artery are decreased during or after a bout of uninterrupted sitting. A bout of prolonged sitting also causes blood pressure and fluctuations in blood pressure to increase. Importantly, we reported that fluctuations in blood pressure caused by sitting are higher in young males versus females, but average blood pressure was higher among females. These findings suggest that sitting exerts sex differences in the control of blood pressure. Importantly, these effects were only demonstrated during the 2-hour bout of sitting. As such, it is unknown whether blood pressure is negatively impacted after prolonged sitting. The proposed study will determine the impact of EDHFs on blood pressure regulation following a 2-hour bout of prolonged sitting among a group of healthy males and females. Continuous heart rate (via electrocardiogram) and blood pressure (via finger cuff), as well as blood flow from the common carotid artery (in the neck), middle cerebral artery (in the brain) and popliteal artery (behind the knee) will be measured before and after sitting (via ultrasound). The ability of the popliteal artery to relax will be assessed using ultrasound following the release of a pressure cuff. Finally, 24-hour blood pressure and heart rate will be recorded after sitting using a monitor worn for 24-hours. The role of EDHFs will be investigated by comparing 1) baseline blood flow and blood pressure responses (no sitting), 2) blood pressure responses following a 2-hour bout of sitting, and 3) the blood pressure responses following a 2-hour bout of sitting while suppressing the release of EDHFs (via fluconazole ingestion).

ELIGIBILITY:
Inclusion Criteria:

* Are between the ages of 18-65.
* Have a body mass index of <40kg/m2 (non-obese).
* Have not smoked nicotine or marijuana-containing products most days of the week within the past 6 months.
* Have not been diagnosed with a cardiovascular, cerebrovascular, respiratory, or metabolic disease.
* Are normotensive.
* Are not currently taking any medications for cardiovascular, metabolic, pulmonary, or neurological disorders, or taking sildenafil regularly.
* Are not allergic to the adhesive used to secure the activPAL activity monitors.
* Are not pregnant or breastfeeding.
* Are not regularly taking any of the following: another anti-fungal, heartburn medications containing cisapride (e.g., Propulsid), depression medications containing amitriptyline (e.g., Elavil) or nortriptyline (e.g., Pamelor), erythromycin (antibiotic), lipid lower medications (i.e., statins), non-steroidal anti-inflammatory drugs (e.g., ibuprofen), or vitamin A supplements.

Exclusion Criteria:

* o Younger than 18 years old. Individuals younger than 18 demonstrate more variable peak FMD responses and require multiple assessments to determine peak response.

  * Over the age of 65. There are age-related impacts on arterial function and the responses to sitting.
  * Body mass index of >40 kg/m2 (i.e., obese II category)(6-8).
  * Smoked nicotine or marijuana-containing products most days of the week within the past 6 months. Cardiovascular health for participants who smoke is poor compared to those who do not smoke, which will negatively impact our arterial function outcomes.
  * Have been diagnosed with a cardiovascular, cerebrovascular, respiratory, or metabolic disease. Such conditions impact our assessments of arterial health. The results of unhealthy participants are not of interest in this study.
  * Hypertension (seated resting systolic pressure >139 mmHg and/or diastolic pressure >89 mmHg). Hypertensive individuals have impairments in artery health, which will affect their baseline artery health measures.
  * Hypotensive (seated resting systolic pressure <90 mmHg and/or diastolic pressure <60 mmHg). Hypotensive people are more likely to experience further reductions in blood pressure during the sitting protocol, which will increase the risk of fainting and/or dizziness.
  * Have a history of fainting and/or dizziness during sitting or standing.
  * Prescribed medications for cardiovascular, metabolic, pulmonary, or neurological disorders. This includes people using hormone replacement therapy. These medications will interfere with our assessments and interpretation of arterial health.
  * Have a known allergy to the clear medical adhesive used to secure the activPAL activity monitors.
  * Females who are pregnant or breastfeeding. Pregnant and breastfeeding females are ineligible to participate. This is due to the known increases in arterial vasodilation associated with pregnancy related sex hormones.
  * Currently or recently (within the past 6 months) regularly taking sildenafil or other medications that increase the relaxing effects of nitric oxide in arteries. Such medication will influence artery blood flow and flow-mediated dilation responses.
  * Are regularly taking any of the following: another anti-fungal, heartburn medications containing cisapride (e.g., Propulsid), depression medications containing amitriptyline (e.g., Elavil) or nortriptyline (e.g., Pamelor), erythromycin (antibiotic), lipid lower medications (i.e., statins), non-steroidal anti-inflammatory drugs (e.g., ibuprofen), or vitamin A supplements. These are to minimize the chance of a participant experiencing an adverse reaction to the fluconazole tablet.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Popliteal Low-Flow Mediated Constriction | Before prolonged sitting, after 1-hour of sitting, after 2-hours of sitting
  During a period of distal cuff-induced ischemia, the endothelial-dependent vasoconstrictor response will be assessed via Duplex ultrasonography. The popliteal artery will be imaged slightly above the popliteal fossa. The L-FMC response will be quantified as the percent reduction in arterial diameter from baseline to the nadir diameter from the last 30-s of a 5-min distal cuff occlusion period.
Acute Blood Pressure | Before prolonged sitting, after 1-hour of sitting, after 2-hours of sitting.
  Beat-by-beat systolic (SBP) and diastolic (DBP) blood pressure will be measured using finger photoplethysmography for 20 minutes before the bout of prolonged sitting, 20 minutes after 1-hour of sitting, and 20 minutes after 2-hours of sitting. Mean arterial pressure will be quantified as 1/3 SBP + 2/3 DBP.
Ambulatory Blood Pressure | This will be worn for a 24-hour period before the first prolonged sitting session, and for 24-hours after each bout of prolonged sitting.
  Using an ABPMpro Ambulatory Blood Pressure Monitors, habitual blood pressure will be measured every 20-minutes during waking hours, and every 30-minutes during sleeping hours.

SECONDARY OUTCOMES:
Carotid Artery Blood Flow Velocity | Before prolonged sitting, after 1-hour of sitting, after 2-hours of sitting.
  Blood flow velocity will be measured immediately prior to the bifurcation in the common carotid artery using Duplex ultrasonography for 5 minutes.
Middle Cerebral Artery Velocity | Before prolonged sitting, after 1-hour of sitting, after 2-hours of sitting.
  Blood flow velocity will be measured via transcranial Doppler over the trans-temporal window for 5 minutes.
Popliteal Flow Mediated Dilation (FMD) | Before prolonged sitting, after 1-hour of sitting, after 2-hours of sitting.
  Following a period of distal cuff induced ischemia, the endothelial-dependent vasodilator response will be assessed via Duplex ultrasonography. The popliteal artery will be imaged slightly above the popliteal fossa. The FMD response will be quantified as the percent increase in arterial diameter from baseline to the peak diameter following the release of the distal cuff.
Physical Activity Behaviour Questionnaire | At time of study enrolment
  A subjective questionnaire that provides information regarding habitual physical activity and sedentary behaviours.
Heart Rate Variability (HRV) | Acute: Before prolonged sitting, after 1-hour of sitting, after 2-hours of sitting. Ambulatory: 24-hours at baseline, 24-hours after each bout of prolonged sitting.
  Heart rate will be determined using cardiac intervals from a lead II electrocardiography during prolonged sitting, and from the built-in electrocardiogram in the ambulatory blood pressure monitor. HRV will be derived from these waveforms using an offline HRV analysis module. Time-domain (I.e., RMSSD), frequency-domain, low frequency (LF) power, high frequency (HF) power, and the LF/HF ratio will be quantified for each participant.
Carotid Intima Media Thickness (cIMT) | Before prolonged sitting, after 1-hour of sitting, after 2-hours of sitting.
  cIMT will be determined from a 5-minute recording of the carotid artery, imaged prior to the bifurcation using Duplex ultrasonography.
Carotid Artery Distensibility | Before prolonged sitting, after 1-hour of sitting, after 2-hours of sitting.
  Distensibility will be determined from 5-minutes of recorded carotid artery imaging via Duplex ultrasonography, and will be calculated as the difference between average arterial diameter during systole and diastole.
Blood Pressure Varibility (BPV) | Acute: Before prolonged sitting, after 1-hour of sitting, after 2-hours of sitting. Ambulatory: 24-hours at baseline, 24-hours after each bout of prolonged sitting.
  Beat-by-beat BPV during sitting will be quantified using the blood pressure measurements derived from finger photoplethysmography. This will be calculated as the average absolute difference between successive finger blood pressure measurements, for systolic blood pressure, diastolic blood pressure, and mean arterial pressure. Ambulatory BPV will be quantified from the 24-hour blood pressure monitors.
Cardiovagal Baroreflex Sensitivity (cvBRS) | Before prolonged sitting, after 1 hour of sitting, after 2-hours of sitting.
  cvBRS will be quantified from beat-by-beat systolic blood pressure (SBP) and R-R intervals in a cvBRS software. cvBRS outcomes will be quantified from a minimum of 3 sequences in which beat-by-beat SBP changes were ≥1 mmHg and changes in R-R interval were ≥ 1 ms. Overall cvBRS is represented by the average slope of SBP and R-R interval regressions for the pooled sequences, and reported separately for both up and down sequences. Baroreflex effectiveness index (BEI) will be measured as the ratio of the number of SBP ramp-induced changes in RR interval to the total number of SBP ramps observed. This will be reported separately for both up and down sequences. This will be measured over a 20-minute time period.
Habitual Activity & Postures | Before first bout of sitting, after each bout of sitting.
  Habitual activity and postures will be measured using activPAL inclinometer-accelerometers positioned on the torso, thigh, and calf. Monitors will be waterproofed and attached 24-hr/day for 8 days via clear medical adhesive. Physical activity (step counts, physical activity intensity), upright posture and detailed sedentary postures (e.g., sitting versus lying time) will be determined via validated, custom software that was developed and openly published by our group.
Baseline Arterial Diameters | Before prolonged sitting, after 1-hour of sitting, after 2-hours of sitting.
  Arterial diameter of the popliteal and carotid arteries will be determined via Duplex ultrasonography over a minimum of 2-minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Myles W O'Brien, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Dalhousie University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to maintain privacy and confidentiality of the participants.

REFERENCES:
- [Background] Turner JR, Viera AJ, Shimbo D. Ambulatory blood pressure monitoring in clinical practice: a review. Am J Med. 2015 Jan;128(1):14-20. doi: 10.1016/j.amjmed.2014.07.021. Epub 2014 Aug 12. PMID 25107387
- [Background] Pellerine LP, Miller K, Frayne RJ, O'Brien MW. Characterizing objective and self-report habitual physical activity and sedentary time in outpatients with an acquired brain injury. Sports Med Health Sci. 2024 Feb 10;6(4):338-343. doi: 10.1016/j.smhs.2024.02.001. eCollection 2024 Dec. PMID 39309460
- [Background] Bays HE, Toth PP, Kris-Etherton PM, Abate N, Aronne LJ, Brown WV, Gonzalez-Campoy JM, Jones SR, Kumar R, La Forge R, Samuel VT. Obesity, adiposity, and dyslipidemia: a consensus statement from the National Lipid Association. J Clin Lipidol. 2013 Jul-Aug;7(4):304-83. doi: 10.1016/j.jacl.2013.04.001. Epub 2013 May 31. PMID 23890517
- [Background] O'Brien MW, Johns JA, Al-Hinnawi A, Kimmerly DS. Popliteal flow-mediated dilatory responses to an acute bout of prolonged sitting between earlier and later phases of natural menstrual and oral contraceptive pill cycles. J Appl Physiol (1985). 2020 Oct 1;129(4):637-645. doi: 10.1152/japplphysiol.00424.2020. Epub 2020 Aug 13. PMID 32790597
- [Background] Liu H, O'Brien MW, Wu Y, Bustamante CM, Kimmerly DS. An acute bout of prolonged sitting blunts popliteal endothelium-independent dilation in young, healthy adults. J Appl Physiol (1985). 2023 Mar 1;134(3):521-528. doi: 10.1152/japplphysiol.00712.2022. Epub 2023 Jan 19. PMID 36656984
- [Background] Ishikura F, Beppu S, Hamada T, Khandheria BK, Seward JB, Nehra A. Effects of sildenafil citrate (Viagra) combined with nitrate on the heart. Circulation. 2000 Nov 14;102(20):2516-21. doi: 10.1161/01.cir.102.20.2516. PMID 11076826
- [Background] Lopes van Balen VA, van Gansewinkel TAG, de Haas S, van Kuijk SMJ, van Drongelen J, Ghossein-Doha C, Spaanderman MEA. Physiological adaptation of endothelial function to pregnancy: systematic review and meta-analysis. Ultrasound Obstet Gynecol. 2017 Dec;50(6):697-708. doi: 10.1002/uog.17431. PMID 28170124
- [Background] Puranik R, Celermajer DS. Smoking and endothelial function. Prog Cardiovasc Dis. 2003 May-Jun;45(6):443-58. doi: 10.1053/pcad.2003.YPCAD13. PMID 12800127
- [Background] Jarvisalo MJ, Ronnemaa T, Volanen I, Kaitosaari T, Kallio K, Hartiala JJ, Irjala K, Viikari JS, Simell O, Raitakari OT. Brachial artery dilatation responses in healthy children and adolescents. Am J Physiol Heart Circ Physiol. 2002 Jan;282(1):H87-92. doi: 10.1152/ajpheart.2002.282.1.H87. PMID 11748051
- [Background] Tomiyama AJ, Hunger JM, Nguyen-Cuu J, Wells C. Misclassification of cardiometabolic health when using body mass index categories in NHANES 2005-2012. Int J Obes (Lond). 2016 May;40(5):883-6. doi: 10.1038/ijo.2016.17. Epub 2016 Feb 4. PMID 26841729
- [Background] Seals DR, Jablonski KL, Donato AJ. Aging and vascular endothelial function in humans. Clin Sci (Lond). 2011 May;120(9):357-75. doi: 10.1042/CS20100476. PMID 21244363
- [Background] Paterson C, Fryer S, Stone K, Zieff G, Turner L, Stoner L. The Effects of Acute Exposure to Prolonged Sitting, with and Without Interruption, on Peripheral Blood Pressure Among Adults: A Systematic Review and Meta-Analysis. Sports Med. 2022 Jun;52(6):1369-1383. doi: 10.1007/s40279-021-01614-7. Epub 2021 Dec 21. PMID 34932203
- [Background] Petterson JL, O'Brien MW, Johns JA, Chiasson J, Kimmerly DS. Influence of prostaglandins and endothelial-derived hyperpolarizing factors on brachial and popliteal endothelial-dependent function in young adults. J Appl Physiol (1985). 2021 Jan 1;130(1):17-25. doi: 10.1152/japplphysiol.00698.2020. Epub 2020 Oct 29. PMID 33119467
- [Background] Hall JE. Integration and regulation of cardiovascular function. Am J Physiol. 1999 Dec;277(6 Pt 2):S174-86. doi: 10.1152/advances.1999.277.6.S174. PMID 10644245
- [Background] Tremblay MS, Aubert S, Barnes JD, Saunders TJ, Carson V, Latimer-Cheung AE, Chastin SFM, Altenburg TM, Chinapaw MJM; SBRN Terminology Consensus Project Participants. Sedentary Behavior Research Network (SBRN) - Terminology Consensus Project process and outcome. Int J Behav Nutr Phys Act. 2017 Jun 10;14(1):75. doi: 10.1186/s12966-017-0525-8. PMID 28599680
- [Background] Sedentary Behaviour Research Network. Letter to the editor: standardized use of the terms "sedentary" and "sedentary behaviours". Appl Physiol Nutr Metab. 2012 Jun;37(3):540-2. doi: 10.1139/h2012-024. Epub 2012 Apr 27. No abstract available. PMID 22540258
- [Background] Herman KM, Saunders TJ. Sedentary behaviours among adults across Canada. Can J Public Health. 2016 Dec 27;107(4-5):e438-e446. doi: 10.17269/cjph.107.5587. PMID 28026711
- [Background] Waghorn J, Liu H, Wu Y, Rayner SE, Kimmerly DS, O'Brien MW. A Single Bout of Prolonged Sitting Augments Very Short-Term Blood Pressure Variability. Am J Hypertens. 2024 Aug 14;37(9):700-707. doi: 10.1093/ajh/hpae055. PMID 38703068